CLINICAL TRIAL: NCT00325988
Title: NINDS Biomarkers in Multiple Sclerosis Study (BioMS)
Brief Title: Biomarkers in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050063; 05-N-0063
Record Dates: First submitted 2006-05-15; First posted 2006-05-15 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-02-03

CONDITIONS: Multiple Sclerosis
Keywords: Neuroimmunology; Demyelinating Disease; Genetics; Proteins
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases

SUMMARY:
This study will identify biomarkers (genes and proteins) in patients with relapsing-remitting multiple sclerosis (MS) and link them with clinical disease parameters, such as the extent of inflammation and rate of disease progression, to try to better understand the disease. It will examine how the biomarkers may be related to disease development and progression and differences among patients' symptoms and response to treatment.

Patients with relapsing-remitting MS between 18 and 60 years of age who are enrolled in the multi-institutional MS-CombiRx trial may be eligible for this sub-study. Participants have blood tests when they enter the MS-CombiRx study and again after 6 months, 1 year, and 3 years for analysis for genetic and protein analysis.

DETAILED DESCRIPTION:
OBJECTIVE: To identify biomarkers (by gene- and protein expression profiling, single nucleotide polymorphism (SNP) haplotype determination, HLA typing) and link these with clinical- and MRI phenotypes in a large cohort of relapsing-remitting (RR-) MS patients. To identify biomarkers that separate MS patients and healthy, matched controls.

STUDY POPULATION: Up to 1000 patients who are enrolled in and treated under a multi-center trial of combination therapy (MS-CombiRx) using two approved disease-modifying therapies (interferon-beta, IFN-b, Avonex; glatiramer-acetate, GA) as single treatments or in combination. 200 healthy, matched control individuals.

DESIGN: Samples of serum and white blood cells will be obtained on each patient prior to randomization in the MS-CombiRx study and then at 6 months 1, and 3 years following randomization. Samples will be analyzed for SNP haplotype, gene and protein expression, and HLA haplotype. Samples from controls will be analyzed in the same fashion, however, only one time point will be analyzed, and there will be no treatment of controls.

OUTCOME MEASURES: The results of the biomarker studies will be assessed in relationship to both the clinical and MRI phenotype at baseline and to change in disability, relapse rate, response to therapy and change in MRI measures of disease during the 3-year treatment period. Each of the biomarker study components will be analyzed with respect to biomarkers that discriminate between MS patients and controls.

SIGNIFICANCE: Similar to rheumatoid arthritis or autoimmune diabetes multiple sclerosis (MS) is considered a complex disease with autoimmune pathogenesis as well as vulnerability of the target tissue, i.e. the central nervous system (CNS). The results of the biomarker study should provide a better understanding of the disease pathogenesis, of the inter-individual disease heterogeneity, and finally identify biomarkers such as gene- and protein expression signatures and individual genes and proteins that are correlated with responsiveness or non-responsiveness to single drug treatment or the combination of the two drugs. The three years duration of the combination therapy trial will further allow us to gather information on the longitudinal evolution of the identified biomarkers under treatment of MS.

ELIGIBILITY:
* INCLUSION CRITERIA - PATIENTS:

To be eligible for entry into this study, candidates must meet the following eligibility criteria at the time of enrollment:

Between the ages of 18 and 60 years, inclusive.

Diagnosis of Relapsing-Remitting MS.

Expanded Disability Status Scale (EDSS) score between 0 and 5.5, inclusive.

At least 2 exacerbations in the prior three years; one exacerbation may utilize the McDonald MRI criteria for dissemination in time (a new Gd-enhancing lesion demonstrated on a scan done at least 3 months following onset of a clinical attack or a new T2 lesion or Gd-enhancing lesions on a follow-up scan after an additional 3 months).

Give written informed consent prior to any testing under this protocol, including screening tests and evaluations that are not considered part of the subject's routine care.

EXCLUSION CRITERIA - PATIENTS:

Candidates will be excluded from study entry if any of the following exclusion criteria exist at the time of screening (prior to randomization):

Prior use of interferon beta or glatiramer acetate.

Acute exacerbation within 30 days of screening.

Steroids for acute exacerbations (greater than 100 mg/day) within 30 days of study entrance or chronic systemic steroid use.

Evidence of progressive MS.

Use of immunosuppressive or chemotherapeutic agents or IVIg.

Inability to perform the MSFC (Time 25-Foot Walk, 9HPT, and PASAT3).

Inability to undergo baseline MRI scan.

History of any significant cardiac, hepatic, pulmonary, or renal disease; immune deficiency; or other medical conditions that would preclude therapy with interferon beta or glatiramer acetate.

Known history of sensitivity to gadopentate dimeglumine or mannitol.

History of a seizure within the 3 months prior to randomization.

History of suicidal ideation or an episode of severe depression within the 3 months prior to randomization.

Abnormal screening blood tests exceeding any of the limits defined below:

Alanine transaminase (ALT) or aspartate transaminase (AST) greater than two times the upper limit of normal (i.e., greater than 2 times the ULN).

Total white blood cell count less than 2,300/mm(3).

Platelet count less than 80,000/mm(3).

Creatinine greater than 2 times the ULN.

Participation in another experimental clinical trial, without formal approval.

Previous participation after randomization in this study.

History of alcohol or drug abuse within the 2 years prior to randomization.

Female subjects who are currently pregnant, breast-feeding, or plan to become pregnant.

For female subjects, unless postmenopausal or surgically sterile, unwillingness to practice effective contraception, as defined by the investigator, during the study. The rhythm method is not to be used as the sole method of contraception.

Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition that is likely to affect the subject's returning for scheduled follow-up visits on schedule (any physical, mental, or social condition, including history of any episode of suicidal ideation or severe depression defined as any episode that required hospitalization within the previous 3 months).

INCLUSION CRITERIA - CONTROLS:

18 to 60 years inclusive.

EXCLUSION CRITERIA - CONTROLS:

Any significant acute or chronic illness, particularly no autoimmune or chronic inflammatory, -infectious disease.

HIV positive.

No treatment with immunomodulatory, immunosuppressive or chemotherapeutic drugs.

Pregnancy.

Nursing mothers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 858 (Actual)
Dates: Start 2004-12-17; Study Completion 2014-02-03

CONTACTS AND LOCATIONS:
Overall Officials: Steven Jacobson, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wynn DR, Rodriguez M, O'Fallon WM, Kurland LT. A reappraisal of the epidemiology of multiple sclerosis in Olmsted County, Minnesota. Neurology. 1990 May;40(5):780-6. doi: 10.1212/wnl.40.5.780. PMID 2082944
- [Background] Noseworthy JH, Lucchinetti C, Rodriguez M, Weinshenker BG. Multiple sclerosis. N Engl J Med. 2000 Sep 28;343(13):938-52. doi: 10.1056/NEJM200009283431307. No abstract available. PMID 11006371
- [Background] Lublin FD, Reingold SC. Defining the clinical course of multiple sclerosis: results of an international survey. National Multiple Sclerosis Society (USA) Advisory Committee on Clinical Trials of New Agents in Multiple Sclerosis. Neurology. 1996 Apr;46(4):907-11. doi: 10.1212/wnl.46.4.907. PMID 8780061